CLINICAL TRIAL: NCT02706509
Title: Comparison Between the Analgesic Affects of Tramadol® and "Verbal Anesthesia" on Pain Management Associated With the Insertion of Jaydess® in Nulliparous Women
Brief Title: Pain Management Associated With the Insertion of Jaydess® in Nulliparous Women
Acronym: Jaydess
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 0063-15-MMC
Record Dates: First submitted 2016-02-17; First posted 2016-03-11 (Estimated); Last update posted 2016-03-11 (Estimated); Status verified 2016-02

CONDITIONS: IUD Insertion Complication
MeSH Terms: interventions — Tramadol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- oral tramadol (Active Comparator): Patients will receive oral Tramadol 50 mg capsules (n=50)' . After an hour, Jaydess intrauterine device will be inserted.
  Interventions: Drug: Tramadol; Device: Jaydess
- verbal anesthesia (Sham Comparator): 'verbal anesthesia' (n=50) After an hour, Jaydess intrauterine device will be inserted
  Interventions: Behavioral: Verbal anesthesia; Device: Jaydess

INTERVENTIONS:
Drug: Tramadol — patient will receive oral Tramadol 50 mg an hour before IUD insertion
  Other Names: ultram
  Arms: oral tramadol
Behavioral: Verbal anesthesia — patient will receive full explanation about the procedure for five minutes before IUD insertion
  Arms: verbal anesthesia
Device: Jaydess — Patient will go through an insertion of Jaydess intrauterine device.

SUMMARY:
A multicenter prospective interventional comparative study that investigate pain management during Jaydess insertion in nulliparous women that will be tested by the analgesic affects of oral tramadol or 'verbal anesthesia' on the patients.

DETAILED DESCRIPTION:
Most intrauterine contraception (IUC) insertions do not require pain management. However, small proportions of nulliparous women experience substantial pain that needs to be proactively managed No prophylactic pharmacological intervention has been adequately evaluated to support routine use for pain reduction during or after IUC insertion. Women's anxiety about the procedure may contribute to higher levels of perceived pain, which highlights the importance of counselling, and creating a trustworthy, unhurried and professional atmosphere in which the experience of the provider also has a major role; a situation frequently referred to as 'verbal anaesthesia'.

It has been proven in the past that the use of oral Tramadol can reduce the pain in the insertion.

In the study investigators will compare the analgesic affects of oral Tramadol and verbal anesthesia on pain relief during Jaydess insertion in nulliparous women.

ELIGIBILITY:
Inclusion Criteria:

* Nulliparous women aged 18-48 years, interested in a long acting, reversible contraception method. Each read and signed the informed consent.

Exclusion Criteria:

Women suffering from:

* Acute or recurrent pelvic inflammatory disease.
* Acute cervicitis or acute Vaginitis.
* Current cervical intraepithelial lesion.
* Current any genital malignancy.
* Progesterone hypersensitivity.
* progesterone-sensitive tumours (e.g. breast tumours).
* Abnormal vaginal bleeding.
* Congenital or acquired uterine anomaly.
* Distorted uterine cavity e.g. fibroid or polyp.
* Impaired liver functions, or liver tumour.
* Known hypersensitivity to the active substance or to any of the excipients of Jaydess.
* Contraindications to Tramadol according to approved product information:

  * In hypersensitivity to tramadol or any of the excipients.
  * In patients who are receiving monoamine oxidase inhibitors or within 2 weeks (14 days) of their withdrawal.
  * In patients with epilepsy not adequately controlled by treatment.
* Vaginismus.

Ages: 18 Years to 48 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-03; Primary Completion 2017-09 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Evaluation of pre-insertion therapy (oral analgesia and oral Tramadol) as pain management during insertion of Jaydess measured on a VAS (0-100 mm). | Day of insertion
  The primary outcome will be the patient evaluation of pain during the procedure. The patient will be asked to assess the pain according to VAS scale (10-100 mm) 10 minutes after the insertion of Jaydess intrauterine device.

SECONDARY OUTCOMES:
Evaluation of pain during menstruation one month after the insertion of Jaydess intrauterine device | one month after insertion
  The patient will be asked to asses the severity of pain during menstruation one month after the insertion of Jaydess intrauterine device according to VAS scale (1-100 mm)
Evaluation of pain during menstruation six month after the insertion of Jaydess | six month after insertion
  The patient will be asked to asses the severity of pain during menstruation six month after the insertion of Jaydess intrauterine device according to VAS scale (1-100 mm)
Evaluation of the amount of bleeding during menstruation one month after the insertion of Jaydess intrauterine device | one month after insertion
  The patient will be asked to asses the amount of bleeding during menstruation one month after the insertion of Jaydess intrauterine device according to a verbal scale (non, minor, medium, sever, very sever)
Evaluation of the amount of bleeding during menstruation six month after the insertion of Jaydess intrauterine device | six month after insertion
  The patient will be asked to asses the amount of bleeding during menstruation six month after the insertion of Jaydess intrauterine device according to a verbal scale (non, minor, medium, sever, very sever)

IPD SHARING:
Plan to Share IPD: No